CLINICAL TRIAL: NCT03295383
Title: Randomized Double Blind Double Dummy Control Trial Comparing the Safety and Efficacy of Rituximab Versus Oral Cyclophosphamide in Severe Forms of Mucous Membrane Pemphigoid
Brief Title: Randomized Clinical Trial Comparing the Safety and Efficacy of Rituximab Versus Oral Cyclophosphamide in Severe Forms of Mucous Membrane Pemphigoid
Acronym: RITUX-MMP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015/208/HP
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Severe Forms of Mucous Membrane Pemphigoid
Keywords: cyclophosphamide; Rituximab
MeSH Terms: interventions — Rituximab; Cyclophosphamide; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rituximab treatment (Experimental): Rituximab at a dose of 1000 mg (or matching placebo) will be administered by IV infusion on Day 1 and Day 15 whatever the patient's weight, with repeat maintenance rituximab (or matching placebo) administration on Day 182 and Day 197
  cyclophosphamide placebo will be administered orally once daily
  Interventions: Drug: Rituximab 1g IV; Drug: Placebo Oral Tablet
- Cyclophosphamide treatment (Active Comparator): cyclophosphamide will be administered orally once daily at the following initial doses:
  patients younger than 75 years: 1.5 mg/kg/day, orally. patients older than 75 years: 1 mg/kg/day, orally.
  Rituximab placebo (NaCl 0.9 %) will be administered by IV infusion on Day 1 and Day 15 whatever the patient's weight, with repeat maintenance rituximab (or matching placebo) administration on Day 182 and Day 197
  Interventions: Drug: Cyclophosphamide 50Mg Oral Tablet; Drug: Placebo of Rituximab

INTERVENTIONS:
Drug: Rituximab 1g IV — Rituximab at a dose of 1000 mg will be administered by IV infusion on Day 1 and Day 15 whatever the patient's weight, with repeat maintenance rituximab (or matching placebo) administration on Day 182 and Day 197
  Arms: Rituximab treatment
Drug: Cyclophosphamide 50Mg Oral Tablet — cyclophosphamide will be administered orally once daily at the following initial doses:
  * patients younger than 75 years: 1.5 mg/kg/day, orally.
  * patients older than 75 years: 1 mg/kg/day, orally.
  Arms: Cyclophosphamide treatment
Drug: Placebo of Rituximab — Rituximab placebo will be administered by IV infusion on Day 1 and Day 15 whatever the patient's weight, with repeat maintenance rituximab administration on Day 182 and Day 197
  Arms: Cyclophosphamide treatment
Drug: Placebo Oral Tablet — cyclophosphamide placebo will be administered orally once daily
  Arms: Rituximab treatment

SUMMARY:
Mucous membrane pemphigoid (MMP) describes a group of chronic auto-immune bullous diseases (AIBD) of the basement membrane zone (BMZ), characterized by predominant or exclusive mucosal involvement, including oral, naso-pharyngeal, laryngo-tracheal, genital, oesophageal, anal and ocular mucous membranes. Circulating autoantibodies are directed against various antigens of the BMZ: BP180, laminin 332 and type 7 collagen. MMP is a rare disease with an incidence of 1.8 new cases/million inhabitants/year in France.

Scar formation which is secondary to initial inflammation, is a characteristic feature of MMP, leading to major disability (e.g blindness and oesophageal, anal, vaginal stenosis) and life-threatening situations (e.g. laryngeal stenosis leading to respiratory failure).

Dapsone is the first line treatment of mild/moderate forms of MMP. Dapsone is used both as initial treatment, and as maintenance therapy. However, severe forms of MMP can rapidly worsen leading to blindness, aphagia due to esophageal stenosis, respiratory failure due to tracheal or laryngeal stenosis, and urinary and sexual dysfunctions due to genital involvement. These patients are usually treated using immunosuppressive drugs. Indeed, corticosteroids (CS) are not recommended in MMP.

Cyclophosphamide was considered as the most effective immunosuppressant in severe forms of MMP, before the use of rituximab, an anti-CD20 monoclonal antibody (MAb).

Two series from our group have assessed the advantages and disadvantages of IV pulse and oral administration of cyclophosphamide in MMP. Oral administration seems more rapidly effective with 54% of complete remission (CR) after a median time of 24 weeks (16-52 weeks).

The results of 41 patients with severe types of MMP (including a French series of 20 patients) treated with rituximab have been published. Rate of CR after one and two cycles were 66% and 90%, respectively. Clinical improvement was rapid, since a decrease in disease activity was observed after 4 weeks of treatment in 64% of patients.

Our results and those of the literature suggest that rituximab might be more effective than cyclophosphamide, which has been considered as the gold standard of treatment in severe forms of disease, up to now.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥18 years old and ≤ 80 years old with a newly diagnosed or previously diagnosed severe MMP diagnosed according to the International MMP Consensus (Chan 2002) on the following criteria:

   Clinical features: Blisters or erosions predominantly affecting any or all mucous membranes (oral, nasal, pharyngeal, laryngeal, anal, genital, or esophageal,) with or without clinically observable scarring. Ocular involvement includes conjunctival inflammation, shortening of fornices, symblepharon, ankyloblepharon, entropion, trichiasis and corneal neovascularisation.

   Patients with skin involvement must not have more than 2 out of the 4 clinical criteria for bullous pemphigoid (BP) proposed by the French group (Vaillant L et al,1998; Joly P et al. 2004) Direct Immunofluorescence (DIF): Linear deposits of IgG, IgA and/or C3 on the BMZ by DIF of patient's skin or mucous membrane Histology: Sub epithelial blister with or without significant leukocyte infiltrate by standard histology of skin or mucosal lesions, when the skin or mucosal biopsy is possible and appropriate.
2. MMP is defined as "severe" in patients with:

   Sight-threatening ocular disease, and/or Potentially life-threatening laryngeal, tracheal or oesophageal stenosis, and/or Involvement of a mucosal site where there is a risk of scarring stenosis (larynx, trachea, esophagus, anus, foreskin, vagina…) and/or More than one mucosal site involved and/or Mucosal involvement (including exclusive but severe oral involvement defined as an oral MMP DAI score > 10), and/or Skin involvement, which have not achieved control of disease activity despite a one month treatment with dapsone at the maximum dose tolerated or for patients with sight-threatening ocular disease, and/or potentially life-threatening laryngeal, tracheal or oesophageal stenosis, without previous treatment by dapsone
3. Patient having read and understood the information letter and signed the Informed Consent Form
4. Patient with updated vaccinations. It is recommended that a patient's vaccination record and the need for immunization prior to study entry be carefully investigated.
5. For women who are not postmenopausal (≥12 months of non-therapy-induced amenorrhoea) or surgically sterile (absence of ovaries and/or uterus) and who do not plan on having children anymore: agreement to remain abstinent or use two adequate methods of contraception, including at least one method with a failure rate of <1% per year, during the treatment period and for at least 12 months after the last dose of study treatment.

   Abstinence is acceptable only if it is in line with the preferred and usual lifestyle of the patient.

   Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

   Barrier methods must always be supplemented with the use of a spermicide.

   For men: Surgical sterility or agreement to remain abstinent or use a condom during the treatment period and for at least 12 months after the last dose of study treatment and agreement to refrain from donating sperm during this same period.

   Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the patient.

   Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
6. Patient agreement to avoid excessive exposure to sunlight during study participation
7. Patient able to comply with the study protocol, in the investigator's judgment
8. Patient affiliated with, or beneficiary of a social security category

Exclusion Criteria:

1. Patient < 18 years old or > 80 years old
2. Non-consenting patient or patient who cannot be followed regularly
3. Patients with only MMP sequelae (stenosis, fibrosis, without inflammation or disease activity)
4. Patients with Brunsting Perry pemphigoid and exclusive skin lesions without mucosal involvement
5. Karnofsky index < 50% (see Appendix 3)
6. Unstable angina or advanced ischemic cardiopathy (extensive myocardial infarction within the last 3 months or post-infarction heart failure)
7. Severe heart failure (NYHA Class III or IV) or severe uncontrolled cardiac disease
8. Uncontrolled cardiac rhythm disorders
9. Severe bronchial obstruction
10. Past history of malignant disease in the previous 10 years, or current progressive malignant disease, except basal cell carcinoma, and squamous cell carcinoma of the skin that have been treated or excised and cured, in situ cervix carcinoma, or any situation in which the oncologist in charge of the patient considers that risk of evolution of severe localisation(s) of MMP is higher than oncologic risk of cyclophosphamide and rituximab.
11. Anemia (haemoglobin < 10 g/ dL ), neutropenia (<1000/mm3), lymphopenia (<900/mm3), thrombopenia (<100 000/mm3)
12. Positive test results for hepatitis B surface antigen (HBsAg), hepatitis B core, antibody (HBcAb), or hepatitis C virus (HCV) serology at screening
13. Liver insufficiency, major renal insufficiency (creatinin clearance ≤ 30 ml/min)
14. Currently active alcohol or drug abuse, or history of alcohol or drug abuse within 24 weeks prior to screening
15. Patients with positive blood test for HIV
16. Inherited or acquired severe immune deficiency
17. Known active infection of any kind (excluding fungal infections of nail), or recent episode of infection, which has required oral antibiotic treatment within 2 weeks prior to enrollment in the trial
18. Infection having required hospitalization, or IV antibiotic treatment within 4 weeks prior to enrollment
19. Past history of severe infection such as fasciitis, osteomyelitis septic arthritis during the year prior to enrollment. Entry into this study may be reconsidered once the infection has fully resolved
20. Evidence of any new or uncontrolled concomitant disease that, in the investigator's judgment, would preclude patient participation, including but not limited to nervous system, renal, hepatic, endocrine, malignant, or gastrointestinal disorders
21. Any concomitant condition that required treatment with oral or systemic corticosteroids within 12 weeks prior to randomization
22. Major surgery within 4 weeks prior to randomization, excluding diagnostic surgery.
23. Patients having received immunosuppressive treatment (such as cyclosporine, mycophenolate mofetil, azathioprine), or any other treatment that might potentially be active on MMP lesions (anti-TNF) within 4 weeks prior to baseline.
24. Treatment with intravenous immunoglobulins, plasmapheresis, or other similar procedure within 8 weeks prior to randomization
25. Previous treatment of MMP with one of the test products: cyclophosphamide or rituximab
26. Previous treatment with a B cell-targeted therapy other than rituximab (e.g., anti-CD20, anti-CD22, or anti-BLyS)
27. Treatment with a live or attenuated vaccine within 28 days prior to randomization
28. Contraindication to MABTHERA 500 mg concentrate for solution for infusion
29. Contraindication to ENDOXAN 50 mg, tablets
30. Contraindication to methylprednisolone marketed as 120 mg powder for injectable solution pharmaceutical form
31. Contraindication to paracetamol marketed as 10 mg/ml solution for infusion pharmaceutical form
32. Contraindication to hydroxyzine marketed as 100 mg / 2 ml injectable solution pharmaceutical form
33. Contraindication to sodium chloride marketed as 0,9% sodium chloride solution for infusion pharmaceutical form
34. Contraindication to glucose marketed as 5% glucose solution for infusion pharmaceutical form
35. Lactose intolerance
36. Lack of peripheral venous access
37. Women pregnant or lactating, or intending to become pregnant during and for 12 months following the study. Women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative result from a serum pregnancy test within 1 week prior to randomization.
38. Patients who plan on having children (due to the risk of amenorrhoea/azoospermia related to cyclophosphamide) and due to the long retention time of rituximab in B cells depleted patients, women of childbearing potential should use effective contraceptive methods during and for 12 months following treatment with MABTHERA
39. Participation in another interventional clinical trial within 28 days prior to randomization and during the study
40. Person deprived of liberty by administrative or judicial decision or placed under judicial protection (guardianship or supervision)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2019-07-11 (Actual); Primary Completion 2022-11-02 (Estimated); Study Completion 2023-11-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving CR or Partial Remission (PR) | Month 12
  Complete remission: absence of any inflammatory lesion, blister or erosion, and, absence of new fibrosing lesions, and/or absence of worsening of established fibrosing lesions Partial remission: presence of transient new inflammatory lesions, blisters or erosions that heal within one week without treatment and, absence of new fibrosing lesions, and/or absence of worsening of established fibrosing lesions. (Murrell D et al. 2015)

SECONDARY OUTCOMES:
Mean evolution of MMP DAI activity score | Month 24
  MMP DAI score is a scoring system who include 2 sub scores: the MMP DAI activity score which assesses disease activity (mucous membrane and skin erosions and blisters), and the MMP DAI damage score, which assesses disease damage (mucous membrane and skin scaring and pigmentation). These 2 "activity" and "damage" sub scores enable distinction between active erosions and blisters from post inflammatory changes and scarring from resolving lesions.
Mean evolution of MMP DAI activity score | Month 6
  MMP DAI score is a scoring system who include 2 sub scores: the MMP DAI activity score which assesses disease activity (mucous membrane and skin erosions and blisters), and the MMP DAI damage score, which assesses disease damage (mucous membrane and skin scaring and pigmentation). These 2 "activity" and "damage" sub scores enable distinction between active erosions and blisters from post inflammatory changes and scarring from resolving lesions.
Evolution of MMP DAI activity score | Month 12
  MMP DAI score is a scoring system who include 2 sub scores: the MMP DAI activity score which assesses disease activity (mucous membrane and skin erosions and blisters), and the MMP DAI damage score, which assesses disease damage (mucous membrane and skin scaring and pigmentation). These 2 "activity" and "damage" sub scores enable distinction between active erosions and blisters from post inflammatory changes and scarring from resolving lesions.
Number of flares / relapses | Month 24
  relapse / flare is defined as "the reappearance of at least 3 new lesions a month (blisters, erosions) that do not heal within one week, or the extension of established lesions in a patient who has achieved disease control." (Murrell D et al. 2015).
Evolution of quality of life score (TAB QOL) | Month 12
  ABQOL score is a quality of life questionnaires specifically developed for patients with autoimmune blistering disorders to assess quality of life (ABQOL)
Evolution of quality of life score AB QOL | Month 12
  TAB QOL score is a quality of life questionnaires specifically developed for patients with autoimmune blistering disorders to assess evolution under treatment (TAB QOL)

CONTACTS AND LOCATIONS:
Overall Officials: Pascal JOLY, Pr, Principal Investigator — University Hospital, Rouen
Locations (27):
- France (27):
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CH Argenteuil, Argenteuil
  - CHU Bordeaux, Bordeaux
  - Brest University Hospital, Brest
  - CHU Caen, Caen
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHU Dijon, Dijon
  - CH Le Mans, Le Mans
  - CHU Lille, Lille
  - CHU de Limoges, Limoges
  - HCL, Lyon
  - APHM La Timone, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - APHP Avicennes, Paris
  - APHP Bichat, Paris
  - APHP Cochin, Paris
  - APHP Henri Mondor, Paris
  - APHP Pitié Salpétrière, Paris
  - APHP Saint-Louis, Paris
  - CH Quimper, Quimper
  - CHU de Reims, Reims
  - CHU Rennes, Rennes
  - CHU saint-Etienne, Saint-Etienne
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No